CLINICAL TRIAL: NCT02820038
Title: Enhancing Patient Ability to Understand and Utilize Complex Information Concerning Medication Self-management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The University of Texas at Dallas (Other); University of Alabama at Birmingham (Other); University of Texas Southwestern Medical Center (Other); University of Pittsburgh Medical Center (Other); Global Healthy Living Foundation (Other); Dartmouth College (Other); Cornell University (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Other
Other Study IDs: 15-2972
Record Dates: First submitted 2016-06-27; First posted 2016-06-30 (Estimated); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2019-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Other CMI Only (Active Comparator): Approximately 75 participants will be assigned to this study group. Participants will ONLY receive medication guides, or other comparable Consumer Medication Information (CMI), for rheumatoid arthritis medications.
  Interventions: Behavioral: Medication Guides
- Other CMI & SMART Program (Experimental): Approximately 75 participants will be assigned to this study group. Participants will receive medication guides, or other comparable Consumer Medication Information (CMI), for rheumatoid arthritis medications AND will be enrolled into the Strategic Memory Advanced Reasoning Training (SMART) Program.
  Interventions: Behavioral: Medication Guides; Behavioral: SMART Program
- Drug Facts Boxes Only (Experimental): Approximately 75 participants will be assigned to this study group. Participants will ONLY receive Drug Facts Boxes for rheumatoid arthritis medications.
  Interventions: Behavioral: Drug Facts Boxes
- Drug Facts Boxes & SMART Program (Experimental): Approximately 75 participants will be assigned to this study group. Participants will receive Drug Facts Boxes for rheumatoid arthritis medicationsAND will be enrolled into the Strategic Memory Advanced Reasoning Training (SMART) Program.
  Interventions: Behavioral: SMART Program; Behavioral: Drug Facts Boxes

INTERVENTIONS:
Behavioral: Medication Guides — The investigators will compare the effectiveness of two types of written prescription drug information targeted for patients: (1) Medication Guides mandated by the Food and Drug Administration, and (2) Drug Facts Boxes, developed by Woloshin and Schwartz.
  Arms: Other CMI & SMART Program; Other CMI Only
Behavioral: SMART Program — The investigators will determine if the effectiveness of written medication information can be increased by Gist Reasoning Training, delivered via the SMART Program, which is designed to enhance patients' ability to extract meaningful gist from complex information.
  Arms: Drug Facts Boxes & SMART Program; Other CMI & SMART Program
Behavioral: Drug Facts Boxes — The investigators will compare the effectiveness of two types of written prescription drug information targeted for patients: (1) Medication Guides mandated by the Food and Drug Administration, and (2) Drug Facts Boxes, developed by Woloshin and Schwartz.
  Arms: Drug Facts Boxes & SMART Program; Drug Facts Boxes Only

SUMMARY:
The aim of the proposed project is to compare the effectiveness of two strategies designed to enhance patient understanding of medication risks/benefits: (1) Medication Guides, mandated for many medications by the Food and Drug Administration and (2) Drug Facts Boxes, developed by Woloshin and Schwartz to enhance the usability of consumer medication information. The investigators will also assess whether the effectiveness of these communication strategies can be increased by Gist Reasoning Training, which is designed to enhance patients' ability to extract meaningful gist from complex information.The investigators anticipate enrolling 300 individuals with rheumatoid arthritis. The study will use a randomized controlled trial design with four study arms. Data will be collected primarily via self-administered, Internet-based surveys using REDCap. All participants will be followed for 6 months after the completion of baseline data collection.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic, autoimmune disorder affecting 0.5% to 1% of the adult population in developed countries worldwide. Current guidelines underscore the importance of aggressive treatment of RA with disease modifying antirheumatic drugs (DMARDS) to control inflammation. Aggressive treatment has been shown to improve patient-centered outcomes, including better symptom control, functional status, and health-related quality of life and reduce the risk of premature death. A major issue in implementing aggressive therapy in practice, however, involves patient reluctance to escalate therapy when they believe that their symptoms are tolerable, despite the presence of active disease, due to concerns about medications risks. Moreover, patients often find it difficult to obtain accurate and personally-relevant information about medication risks and benefits that is written in language they can understand. There is a clear gap between the information patients want about medication risks and benefits and the information they currently receive as part of routine care.

The aim of the proposed project is to compare the effectiveness of two strategies designed to enhance patient understanding of medication risks/benefits: (1) Medication Guides, mandated for many medications by the Food and Drug Administration and (2) Drug Facts Boxes, developed by Woloshin and Schwartz to enhance the usability of consumer medication information. The investigators will also assess whether the effectiveness of these communication strategies can be increased by Gist Reasoning Training, which is designed to enhance patients' ability to extract meaningful gist from complex information.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Able to speak and read in English
3. Physician confirmed RA define by 1987 American College of Rheumatology criteria
4. Moderate or highly active rheumatoid arthritis (assess by Routine Assessment of Patient Index Data 3 (RAPID3) score > 2.0) and
5. Physician indicates patient is a candidate for initiation or escalation of Disease-modifying antirheumatic drug (DMARD) therapy

Exclusion Criteria:

1. Hearing or visually impaired

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2016-09; Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Blalock, PhD, Principal Investigator — UNC; Caprice Hunt, MPH, Study Director — UNC
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will create a web-site to disseminate study findings. Access to the website will not be restricted in any way. The website will provide a link for individuals to obtain a copy of study data. Individuals will be required to complete a form to request the data, indicating their name, contact information, and the research questions they plan to address. The investigators will then provide individuals with a complete, cleaned, deidentified copy of the final Statistical Analysis Software (SAS) dataset and a copy of the study protocol which will include all of the information needed to replicate the analyses or perform secondary analyses. The investigators will use SharePoint to provide these materials to those who request them. The link providing access to study data will appear and be active within nine months following the final year of funding. The reason for not putting the data onto the study website is to enable the investigators to track data usage.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All materials will be made available by 2/15/2020 and will remain available via the website for at least two years.
Access Criteria: Completion of a form indicating the name of the requester, contact information, and the research questions the requester plans to address. Completion of this form is only required to ensure that the requester is not a bot.

REFERENCES:
- [Derived] Blalock SJ, Solow EB, Reyna VF, Keebler M, Carpenter D, Hunt C, Hickey G, Curtis JR, O'Neill K, Chapman SB. Enhancing Patient Understanding of Medication Risks and Benefits. Arthritis Care Res (Hoboken). 2022 Jan;74(1):142-150. doi: 10.1002/acr.24421. Epub 2021 Dec 22. PMID 32799397

RESULTS

PARTICIPANT FLOW:
Groups:
- Other CMI Only: Participants were given access to Medication Guides, mandated by the Food and Drug Administration for many medications used to treat rheumatoid arthritis, or comparable consumer medication information for medications without a mandated medication guide.
- Other CMI & SMART Program: Participants were given access to Medication Guides, mandated by the Food and Drug Administration for many medications used to treat rheumatoid arthritis, or comparable consumer medication information for medications without a mandated medication guide.
  Participants were also invited to participate in gist reasoning training, delivered via the SMART Program, which is designed to enhance patients' ability to extract meaningful gist from complex information.
- Drug Facts Boxes Only: Participants were given access to medication information in the Drug Facts Box format developed by Woloshin and Schwartz.
- Drug Facts Boxes & SMART Program: Participants were given access to medication information in the Drug Facts Box format developed by Woloshin and Schwartz.
  Participants were also invited to participate in gist reasoning training, delivered via the SMART Program, which is designed to enhance patients' ability to extract meaningful gist from complex information.
Period: Overall Study
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Started (Numbers are those who completed baseline data collection and given access to intervention materials) | 78 | 77 | 65 | 66
Completed | 68 | 52 | 60 | 44
Not Completed | 10 | 25 | 5 | 22
Not completed — Lost to Follow-up | 7 | 11 | 2 | 9
Not completed — Withdrawal by Subject | 3 | 14 | 3 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program | Total
Number analyzed (Participants) | 78 | 77 | 65 | 66 | 286
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (10.8) | 54.7 (11.8) | 56.2 (10.1) | 54.9 (14.7) | 55.3 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 69 | 60 | 59 | 258
  Male | 8 | 8 | 5 | 7 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 3 | 6 | 17
  Not Hispanic or Latino | 66 | 64 | 54 | 52 | 236
  Unknown or Not Reported | 9 | 8 | 8 | 8 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2 | 1 | 5
  Asian | 2 | 1 | 1 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 10 | 11 | 11 | 44
  White | 58 | 62 | 47 | 47 | 214
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 3 | 4 | 6 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78 | 77 | 65 | 66 | 286
Met Criteria for Informed Decision-Making [Count of Participants; unit: Participants] — Informed decision making involves making a value-consistent decision based on accurate knowledge. Knowledge was assessed as described under Outcome 2. Values were assessed using a scale ranging from 0 to 10, with lower scores reflecting reluctance to use medications. Participants were classified as making an informed choice if they: (1) answered at least 85% of the knowledge items correctly, scored 6 or more on the values scale, and were currently taking a DMARD OR (2) answered 85% of the knowledge items correctly, scored 5 or less on the values measure, and were not taking a DMARD. Population: One participant had missing data on medication use at baseline.
  Participants
    number analyzed (Participants) | 77 | 77 | 65 | 66 | 285
    (all) | 29 | 28 | 25 | 20 | 102

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Classified as Having Made an Informed Decision at 6 Months
Description: Informed decision making is characterized by making a value-consistent decision based on accurate knowledge. Knowledge will be assessed as described under Outcome 2. Values will be assessed using a 10-item scale developed by Fraenkel et al. Scores on this scale can range from 0 to 10, with lower scores reflecting a reluctance to use medications to control disease activity. Participants will be classified as having made an informed choice if they: (1) answered at least 85% of the knowledge items correctly, scored 6 or more on the values scale, and are currently taking one or more DMARDS OR (2) answered 85% of the knowledge items correctly, scored 5 or less on the values measure, and are not currently taking a DMARD. Otherwise, individuals will be classified as not having made an informed choice.
Time Frame: Month 6 Follow-up
Population: Includes 221 participants who had sufficient data to classify as either meeting or not meeting the criteria for informed decision-making at the 6-month follow-up. (Excludes 65 people who had missing data at the 6-month follow-up.)
Measure: Number; unit: percentage of participants
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 67 | 52 | 59 | 43
percentage of participants
  % Not Informed Per Criteria | 59.7 | 44.2 | 49.2 | 55.8
  % Informed Per Criteria | 40.3 | 55.8 | 50.9 | 44.2
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would be more likely to meet the criteria for Informed Decision-Making at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority; p = 0.8408, Regression, Logistic; Regression model adjusted for whether participant met criteria for informed decision making at baseline; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.52 to 2.24] — Modeled probability of meeting criteria for informed decision making at the 6-month follow-up. Independent variable coded: 0=Other Consumer Medication Information (CMI) Only, Other CMI+SMART, DrugFactsBox® (DFB) Only; 1=DFB+SMART
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would be more likely to meet the criteria for Informed Decision-Making at the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority; p = 0.58, Regression, Logistic; Regression model adjusted for whether participant met criteria for informed decision making at baseline; Odds Ratio (OR) = 1.18, 95% CI 2-sided [0.66 to 2.12] — Modeled probability of meeting criteria for informed decision making at the 6-month follow-up. Independent variable coded: 0=Other CMI Only or Other CMI+SMART, 1=DFB or DFB + SMART
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would be more likely to meet the criteria for Informed Decision-Making at the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority; p = 0.1937, Regression, Logistic; Regression model adjusted for whether participant met criteria for informed decision making at baseline; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.82 to 2.68] — Modeled probability of meeting criteria for informed decision making at the 6-month follow-up. Independent variable coded: 0=Other CMI Only or DFB Only, 1=Other CMI + SMART or DFB+SMART
Statistical Analysis 4: Comparison: Other CMI Only vs Drug Facts Boxes Only; In this analysis, participants were restricted to those who did not meet criteria for informed decision-making at baseline; Test type: Superiority; p = 0.0193, Regression, Logistic; Sample restricted to participants who did not meet the criteria for informed decision making at baseline; Odds Ratio (OR) = 2.379, 95% CI 2-sided [1.15 to 4.92] — [estimate comment as in outcome 1, analysis 3]
Statistical Analysis 5: Comparison: Other CMI Only vs Drug Facts Boxes Only; In this analysis, participants were restricted to those who met the criteria for informed decision-making at baseline; Test type: Superiority; p = 0.2216, Regression, Logistic; Odds Ratio (OR) = 0.53, 95% CI 2-sided [0.19 to 1.48] — [estimate comment as in outcome 1, analysis 3]

2. Secondary Outcome: Mean Knowledge of the Risks and Benefits Associated With DMARD Therapy at 6 Months Adjusted for Baseline
Description: Knowledge of DMARD risks and benefits will be assessed by measures developed by Fraenkel et al., Barton et al., and Fayet et al. The combined measure will have a total of 36 items. Most items are answered on a true/false scale (with a don't know option provided). Each correct response will receive 1-point (maximum of 36 points). Scores transformed to a 100-point scale (ranging from 0-100) with higher values reflecting greater knowledge.
Time Frame: Month 6 Follow-up
Population: Includes 223 participants who had sufficient data to classify as either meeting or not meeting the criteria for informed decision-making at the 6-month follow-up. (Excludes 63 people who had missing data at the 6-month follow-up.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 68 | 52 | 59 | 44
score on a scale | 81.9 (0.9) | 84.0 (1.1) | 82.1 (1.0) | 84.4 (1.2)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in knowledge between baseline and the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.1630, Regression, Linear; Mean Difference (Net) = -1.83, 95% CI 2-sided [-1.83 to 0.75], Standard Error of Mean 1.32 — Independent variable coded: 0=Other CMI Only, Other CMI+SMART, DFB Only; 1=DFB+SMART. Difference score calculated as: Comparison Group - Intervention Group. Thus, negative values indicate mean was greater in the intervention group
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in knowledge between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.7892, Regression, Linear; Mean Difference (Net) = -0.28, 95% CI 2-sided [-2.33 to 1.77], Standard Error of Mean 1.05; Independent variable coded: 0=Other CMI Only, DFB Only; 1=DFB+SMART, Other CMI+SMART. Difference score calculated as: Comparison Group - Intervention Group. Thus, negative values indicate mean was greater in the intervention group
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in knowledge between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.0377, Regression, Linear; Mean Difference (Net) = -2.19, 95% CI 2-sided [-4.25 to -0.13], Standard Error of Mean 1.05 — Independent variable coded: 0=Other CMI Only, DFB Only; 1=DFB+SMART, Other CMI+SMART. Difference score calculated as: Comparison Group - Intervention Group. Thus, negative values indicate mean was greater in the intervention group

3. Secondary Outcome: Mean Values at 6-Months Adjusted for Baseline
Description: Values. Questions included in the self-administered questionnaires asked participants to indicate the extent to which they agreed or disagreed with 10 simple values statements (e.g., It is OK to ignore the risk of a serious side effect if it is extremely rare; It is better to continue with the pain I know than to change my medications) developed by Fraenkel and colleagues. Responses were recorded on a 4-point scale ranging from 1=Strongly Agree to 4=Strongly Disagree. Responses were then summed and rescored to yield a composite scale that ranged from -15 to +15, where positive numbers reflected values favoring the use of medications to control rheumatoid arthritis (RA) disease activity.
Time Frame: Month 6 Follow-up
Population: Includes 218 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 68 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Other CMI & SMART Program: Participants were given Medication Guides, mandated by the Food and Drug Administration for many medications used to treat rheumatoid arthritis, or comparable consumer medication information for medications without a mandated medication guide.
  Participants were also invited to participate in gist reasoning training, delivered via the SMART Program, which is designed to enhance patients' ability to extract meaningful gist from complex information.
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 66 | 52 | 58 | 42
score on a scale | 6.3 (0.4) | 5.6 (0.4) | 5.5 (0.4) | 5.8 (0.5)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in values favorable to aggressive therapy between baseline and the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.9216, Regression, Linear; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.98 to 1.08], Standard Error of Mean 0.53; Independent variable coded: 0=Other CMI Only, Other CMI+SMART, DFB Only; 1=DFB+SMART. Difference score calculated as: Comparison Group - Intervention Group. Thus, negative values indicate mean was greater in the intervention group
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in values favoring aggressive therapy between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.3843, Regression, Linear; Mean Difference (Net) = 0.36, 95% CI 2-sided [-0.45 to 1.17], Standard Error of Mean 0.42 — Independent variable coded: 0=Other CMI Only, Other CMI+SMART; 1=DFB Only, DFB+SMART. Difference score calculated as: Comparison Group - Intervention Group. Thus, negative values indicate mean was greater in the intervention group
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in values favoring aggressive therapy between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5090, Regression, Linear; Mean Difference (Net) = 0.27, 95% CI 2-sided [-0.54 to 1.09], Standard Error of Mean 0.42 — [estimate comment as in outcome 2, analysis 3]

4. Secondary Outcome: Mean Gist Reasoning Ability, Lesson Quality at 6 Month Follow-up Adjusted for Baseline
Description: The investigators used the Test of Strategic Learning (TOSL) to quantify participants' ability to abstract gist meanings from complex text. The TOSL consists of 4 text passages varying in length (from 291 to 575 words) and complexity. Each participant responded to one passage at each time point. Participants were asked to provide a summary of the original text, focused on bottom-line-meaning rather than specific details. Responses were scored to assess the quality of high-level interpretations (Lesson Quality, range 0 to 5) using an objective scoring system by a trained and experienced rater, blinded to participants' group assignment and time point of testing. Higher scores reflect better lesson quality.
Time Frame: Month 6 Follow-up
Population: Includes 177 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 109 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 56 | 41 | 48 | 32
score on a scale | 1.1 (0.2) | 0.8 (0.2) | 1.0 (0.2) | 1.3 (0.2)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater increases in gist reasoning ability at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.1486, Regression, Linear; Mean Difference (Net) = -0.33, 95% CI 2-sided [-0.77 to 0.12], Standard Error of Mean 0.23 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in gist reasoning ability between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.4888, Regression, Linear; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.47 to 0.22], Standard Error of Mean 0.18 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in gist reasoning ability between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.8637, Regression, Linear; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.32 to 0.38], Standard Error of Mean 0.18 — [estimate comment as in outcome 2, analysis 3]

5. Secondary Outcome: Mean Gist Reasoning Ability, Complex Abstraction at 6-Month Follow-up Adjusted for Baseline
Description: The investigators used the Test of Strategic Learning (TOSL) to quantify participants' ability to abstract gist meanings from complex text. The TOSL consists of 4 text passages varying in length (from 291 to 575 words) and complexity. Each participant responded to one passage at each time point. Participants were asked to provide a summary of the original text, focused on bottom-line-meaning rather than specific details. Responses were scored to assess the number of abstracted ideas (Complex Abstraction, range 0 to 8) using an objective scoring system by a trained and experienced rater, blinded to participants' group assignment and time point of testing. Higher scores indicate more ideas abstracted.
  The investigators will assess change in the total score over time from baseline to 6 month follow-up.
Time Frame: Month 6 Follow-up
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 56 | 41 | 48 | 32
score on a scale | 2.0 (0.2) | 2.0 (0.2) | 1.9 (0.2) | 1.8 (0.2)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater gist reasoning ability at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5070, Regression, Linear; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.33 to 0.66], Standard Error of Mean 0.25 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; [analysis description as in outcome 4, analysis 2]; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.4821, Regression, Linear; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.25 to 0.52], Standard Error of Mean 0.19 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; [analysis description as in outcome 4, analysis 3]; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.7777, Regression, Linear; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.33 to 0.44], Standard Error of Mean 0.20 — [estimate comment as in outcome 2, analysis 3]

6. Secondary Outcome: Mean Satisfaction With Medication Information at 6-Month Follow-up Adjusted for Baseline
Description: This outcome will be assessed by the 17-item Satisfaction with Information about Medicines Scale (SIMS). Items ask participants to rate the amount of information they have received about different aspects of their medications. Responses are summed across items to yield a total score with a possible range of 0 to 17, with higher scores reflecting greater satisfaction with the amount of information received.
Time Frame: Month 6 Follow-up
Population: Includes 206 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 80 people with missing data.)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 65 | 49 | 55 | 37
score on a scale | 13.0 (0.4) | 12.6 (0.5) | 12.6 (0.5) | 12.4 (0.6)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater increases in satisfaction at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.6084, Regression, Linear; Mean Difference (Net) = 0.33, 95% CI 2-sided [-0.93 to 1.58], Standard Error of Mean 0.64 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in satisfaction between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5970, Regression, Linear; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.71 to 1.23], Standard Error of Mean 0.50 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in satisfaction between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = .5094, Regression, Linear; Mean Difference (Net) = 0.33, 95% CI 2-sided [-0.65 to 1.31], Standard Error of Mean 0.50 — [estimate comment as in outcome 2, analysis 3]

7. Secondary Outcome: Mean Overall Treatment Satisfaction at 6-Month Follow-up Adjusted for Baseline
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM-9) will be used to assess treatment satisfaction. TSQM-9 has 3 subscales: effectiveness, convenience and overall satisfaction. Items ask participants to rate their satisfaction with difference aspect of their treatment regimen on a 7-point scale with endpoints labeled, Extremely Dissatisfied (1) and Extremely Satisfied (7). Internal consistency of each subscale has been demonstrated with Cronbach's alpha exceeding 0.80 for each sub-scale. Each subscale has been shown to discriminate between individuals classified as exhibiting Low vs. Medium medication adherence. The investigators combined items across all three subscales to yield a measure of overall treatment satisfaction (range: 0 to 100, with higher scores reflecting greater satisfaction).
Time Frame: Month 6 Follow-up
Population: Includes 210 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 76 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 67 | 50 | 55 | 38
score on a scale | 69.4 (1.9) | 64.6 (2.1) | 66.0 (2.0) | 68.4 (2.5)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; [analysis description as in outcome 6, analysis 1]; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5866, Regression, Linear; Mean Difference (Net) = -1.48, 95% CI 2-sided [-6.85 to 3.89], Standard Error of Mean 2.74 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; [analysis description as in outcome 6, analysis 2]; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.8689, Regression, Linear; Mean Difference (Net) = 0.35, 95% CI 2-sided [-3.82 to 4.52], Standard Error of Mean 2.13 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; [analysis description as in outcome 6, analysis 3]; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = .4356, Regression, Linear; Mean Difference (Net) = 1.66, 95% CI 2-sided [-2.53 to 5.86], Standard Error of Mean 2.14 — [estimate comment as in outcome 2, analysis 3]

8. Secondary Outcome: Mean Arthritis Self-Efficacy at 6-Month Follow-up Adjusted for Baseline
Description: The investigators will assess confidence in one's ability to manage arthritis symptoms in different situations via the 8-item Arthritis Self-Efficacy Scale (e.g., keep pain from interfering with things participants want to do). Responses are recorded on a 100-point scale with endpoints labeled "Very Uncertain" and "Very Certain". This measure has been widely used in arthritis patient populations for over two decades and has been shown to have excellent psychometric properties, including high internal consistency (Cronbach's alpha generally exceeds 0.90) and sensitivity to change following participation in illness self-management programs. To create a total scale score, the investigators summed participant responses across the items in the scale and divided by the number of items answered. Thus, the scale has a possible range of 0 to 100. Higher scores indicate greater self-efficacy.
Time Frame: Month 6 Follow-up
Population: Includes 202 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 84 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 63 | 50 | 53 | 36
score on a scale | 47.4 (2.0) | 48.4 (2.3) | 49.4 (2.2) | 44.9 (2.7)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater increases in self-efficacy at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.2366, Regression, Linear; Mean Difference (Net) = 3.48, 95% CI 2-sided [-2.30 to 9.26], Standard Error of Mean 2.95
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in self-efficacy between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.8841, Regression, Linear; Mean Difference (Net) = 0.33, 95% CI 2-sided [-4.16 to 4.83], Standard Error of Mean 2.29 — [estimate comment as in outcome 2, analysis 3]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in self-efficacy between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5264, Regression, Linear; Mean Difference (Net) = 1.45, 95% CI 2-sided [-3.05 to 5.95], Standard Error of Mean 2.30 — [estimate comment as in outcome 2, analysis 3]

9. Secondary Outcome: Mean Medication Adherence at 6-Month Follow-up Adjusted for Baseline
Description: Medication Adherence was assessed by a single question that asked: "All things considered, how much of the time do you use your RA medications EXACTLY as directed?" Responses were recorded on a 100-point visual analog scale with endpoints labeled "None of the Time" and "All of the time". Higher values reflect greater medication adherence.
Time Frame: Month 6 Follow-up
Population: Includes 181 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 105 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 62 | 41 | 46 | 32
score on a scale | 92.3 (1.4) | 87.9 (1.7) | 95.5 (1.6) | 92.2 (1.9)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater increases in medication adherence at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.9604, Regression, Linear; Mean Difference (Net) = -0.10, 95% CI 2-sided [-4.40 to 4.18], Standard Error of Mean 2.19 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in adherence between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.0279, Regression, Linear; Mean Difference (Net) = -3.62, 95% CI 2-sided [-6.84 to -0.40], Standard Error of Mean 1.64 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in medication adherence between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.0184, Regression, Linear; Mean Difference (Net) = 3.92, 95% CI 2-sided [0.67 to 7.18], Standard Error of Mean 1.66 — [estimate comment as in outcome 2, analysis 3]

10. Secondary Outcome: Mean Illness Intrusiveness at 6-Month Follow-up Adjusted for Baseline
Description: Illness Intrusiveness will be assessed by the 13-item Illness Intrusiveness Ratings Scale. Items ask respondents to rate the degree to which their "illness and/or its treatment" interferes with aspects of life that are essential for quality of life. Responses will be recorded on a visual analog scale, with endpoints labeled Not Very Much (0) and Very Much (100). The instrument will be scored by summing across all items and dividing by the number of items answered to yield a total score ranging from 0 to 100 where higher values reflect greater illness intrusiveness.
Time Frame: Month 6 Follow-up
Population: Includes 205 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 81 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 66 | 50 | 52 | 37
score on a scale | 49.7 (1.8) | 50.0 (2.1) | 45.5 (2.1) | 45.7 (2.5)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater decreases in illness intrusiveness at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.3056, Regression, Linear; Mean Difference (Net) = 2.79, 95% CI 2-sided [-2.56 to 8.14], Standard Error of Mean 2.73 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater decrease in illness intrusiveness between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.0466, Regression, Linear; Mean Difference (Net) = 4.19, 95% CI 2-sided [0.06 to 8.32], Standard Error of Mean 2.11 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater decrease in illness intrusiveness between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.9106, Regression, Linear; Mean Difference (Net) = -.024, 95% CI 2-sided [-4.38 to 3.90], Standard Error of Mean 2.11 — [estimate comment as in outcome 2, analysis 3]

11. Secondary Outcome: Mean Health Distress at 6-Month Follow-up Adjusted for Baseline
Description: Health Distress will be assessed by the 4-item measure developed by Lorig and colleagues. This measure was adapted from the Medical Outcomes Study health distress scare for use in arthritis populations. The adapted measure has demonstrated high internal consistency (Cronbach's alpha= .87) and responsiveness to change following completion of an arthritis self-management course. Participants will respond to each question on a 6-point scale, ranging from None of the Time (0) to All of the Time (5). Thus, the total score will range from 0 to 5, with higher scores reflecting greater Health Distress.
Time Frame: Month 6 Follow-up
Population: Includes 208 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 78 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 66 | 51 | 55 | 36
score on a scale | 2.2 (0.1) | 2.1 (0.1) | 2.1 (0.1) | 2.4 (0.2)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater decreases in health distress at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.1762, Regression, Linear; Mean Difference (Net) = -0.23, 95% CI 2-sided [-0.57 to 0.10], Standard Error of Mean 0.17 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater decrease in health distress between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.4186, Regression, Linear; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.36 to 0.15], Standard Error of Mean 0.13 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater decrease in health distress between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.8848, Regression, Linear; Mean Difference (Net) = -.02, 95% CI 2-sided [-0.28 to 0.24], Standard Error of Mean 0.13 — [estimate comment as in outcome 2, analysis 3]

12. Secondary Outcome: Mean Global Health Status at 6-Month Follow-up Adjusted for Baseline
Description: This outcome will be assessed by a single-item asking participants to rate their current health on a 5-point scare where 1=Poor, 2=Fair, 3= Good, 4= Very Good, and 5= Excellent. This item is part of the Medical Outcomes Study Core Survey Instrument and responses have been shown to predict mortality and health care utilization as well as multi-item health status measures.
Time Frame: Month 6 Follow-up
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 67 | 51 | 55 | 37
score on a scale | 2.5 (0.1) | 2.5 (0.1) | 2.5 (0.1) | 2.5 (0.1)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater increases in health status at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.6403, Regression, Linear; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.15 to 0.25], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in global health status between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.8766, Regression, Linear; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.14 to 0.16], Standard Error of Mean 0.08 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater improvement in global health status between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.7603, Regression, Linear; Mean Difference (Net) = 0.02, 95% CI 2-sided [-0.13 to 0.18], Standard Error of Mean 0.08 — [estimate comment as in outcome 2, analysis 3]

13. Secondary Outcome: Mean Disease Activity at 6-Month Follow-up Adjusted for Baseline
Description: Disease Activity will be assess using the Routine Assessment of Patient Index Data 3 (RAPID3). This instrument is based on the Multi-Dimensional Health Assessment Questionnaire (MDHAQ), which is adapted from the standard HAQ. The RAPID3 includes the 3 Core Data Set measures of physical function, pain, and patient global estimate. The score for physical function ranges from 0 to 10 and is calculated by adding the ten activities of daily living, each scored from 0 to 3 by the patient and dividing the total raw score by 3. Pain and global estimate of health are measured on a likert scale from 0 to 10. The three 0-10 scores for physical function, pain, and global assessment of health are added together and divided by 3 to create a composite score, ranging from 0 to 10. Higher values reflect greater disease activity.
Time Frame: Month 6 Follow-up
Population: Includes 209 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 77 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 66 | 51 | 55 | 37
score on a scale | 4.3 (0.2) | 4.4 (0.2) | 4.2 (0.2) | 4.2 (0.2)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater decreases in disease activity at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.7093, Regression, Linear; Mean Difference (Net) = 0.10, 95% CI 2-sided [-0.43 to 0.63], Standard Error of Mean 0.27 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater decrease in disease activity between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5941, Regression, Linear; Mean Difference (Net) = 0.11, 95% CI 2-sided [-0.30 to 0.52], Standard Error of Mean 0.21 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater decrease in disease activity between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.9476, Regression, Linear; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.42 to 0.40], Standard Error of Mean 0.21 — [estimate comment as in outcome 2, analysis 3]

14. Secondary Outcome: Mean Depression at 6-Month Follow-up Adjusted for Baseline
Description: Depression will be assessed using the Neuro-QOL (Quality of Life in Neurological Disorders) Version 1 item bank. Raw scores are rescaled to a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. The United States general population is used as the reference group. A higher T-score represents greater depression.Thus, a person who has a T-score of 70 is two SDs above the average level of depression observed in the referenced population.
Time Frame: Month 6 Follow-up
Population: Includes 207 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 79 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 66 | 50 | 54 | 37
score on a scale | 49.7 (0.5) | 50.4 (0.6) | 50.4 (0.6) | 50.2 (0.7)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater decreases in depression at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.9128, Regression, Linear; Mean Difference (Net) = -0.09, 95% CI 2-sided [-1.65 to 1.48], Standard Error of Mean 0.80 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater decrease in depression between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.6312, Regression, Linear; Mean Difference (Net) = -0.29, 95% CI 2-sided [-1.50 to 0.91], Standard Error of Mean 0.62 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater decrease in depression between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5766, Regression, Linear; Mean Difference (Net) = -0.35, 95% CI 2-sided [-1.57 to 0.87], Standard Error of Mean 0.62 — [estimate comment as in outcome 2, analysis 3]

15. Secondary Outcome: Mean Fatigue at 6-Month Follow-up Adjusted for Baseline
Description: Fatigue will be assessed using the Neuro-QOL (Quality of Life in Neurological Disorders) Version 1 item bank. Raw scores are rescaled to a standardized T-score with a mean of 50 and a standard deviation (SD) of 10. The United States general population is used as the reference group. A higher T-score represents greater fatigue.Thus, a person who has a T-score of 70 is two SDs above the average level of fatigue observed in the referenced population.
Time Frame: Month 6 Follow-up
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 65 | 50 | 54 | 37
score on a scale | 53.8 (0.7) | 53.9 (0.8) | 54.3 (0.8) | 55.3 (0.9)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit greater decreases in fatigue at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.2123, Regression, Linear; Mean Difference (Net) = -1.30, 95% CI 2-sided [-3.34 to 0.75], Standard Error of Mean 1.04 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater decrease in fatigue between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.2691, Regression, Linear; Mean Difference (Net) = -0.89, 95% CI 2-sided [-2.48 to 0.70], Standard Error of Mean 0.81 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater decrease in fatigue between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5655, Regression, Linear; Mean Difference (Net) = -0.47, 95% CI 2-sided [-2.06 to 1.13], Standard Error of Mean 0.81 — [estimate comment as in outcome 2, analysis 3]

16. Secondary Outcome: Mean Health Literacy at 6-Month Follow-up Adjusted for Baseline
Description: Health literacy will be assessed via the Newest Vital Sign (NVS). This instrument, which tests literacy skills for both numbers and words, has been validated against a previously validated measure of health literacy (the TOFHLA). Participants are given a specially designed ice cream nutrition label to review and are asked a series of questions about the label. 1-point is given for each correct answer (maximum of 6 points). Scores transformed to a 100-point scale (ranging from 0-100) with higher values reflecting greater health literacy.
Time Frame: Month 6 Follow-up
Population: Includes 203 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 83 people with missing data.)
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 66 | 48 | 51 | 38
score on a scale | 73.9 (2.8) | 75.9 (3.3) | 73.9 (3.2) | 72.0 (3.7)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater increases in health literacy at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.5364, Regression, Linear; Mean Difference (Net) = 2.52, 95% CI 2-sided [-5.51 to 10.55], Standard Error of Mean 4.10 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in health literacy between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.6050, Regression, Linear; Mean Difference (Net) = 1.67, 95% CI 2-sided [-4.68 to 8.01], Standard Error of Mean 3.24 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit a greater increase in health literacy between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.9240, Regression, Linear; Mean Difference (Net) = -0.31, 95% CI 2-sided [-6.66 to 6.05], Standard Error of Mean 3.24 — [estimate comment as in outcome 2, analysis 3]

17. Secondary Outcome: Information Seeking: Participating in BetterChoices, BetterHealth
Description: After the 6 week follow-up interview, all participants were given an opportunity to take part in the BetterChoices, BetterHealth program. To assess information seeking, the investigators tracked whether or not participants enrolled in the class and attended at least one class session. This variable was coded such that: 0=Either did not enroll or did not attend any class sessions, 1=Enrolled and attended at least one class session.
Time Frame: 6 months
Population: Includes 277 participants with non-missing data at baseline and at the 6-month follow-up. (Excludes 9 people with missing data.)
Measure: Count of Participants; unit: Participants
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 75 | 73 | 64 | 65
Participants
  Participated in at least one session | 15 | 10 | 14 | 11
  Did not participate in any sessions | 60 | 63 | 50 | 54
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would be more likely to participate in the BetterChoices, BetterHealth program if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority; p = 0.7871, Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.43 to 1.89] — Modeled probability of attending at least one class session. Independent variable coded: 0=Other CMI Only, Other CMI+SMART, DFB Only; 1=DFB+SMART
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would be more likely to participate in at least one session of the BetterChoices,BetterHealth program if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority; p = 0.5815, Regression, Logistic; Odds Ratio (OR) = 1.189, 95% CI 2-sided [0.643 to 2.198] — Modeled probability of attending at least one class. Independent variable coded: 0=Other CMI Only, Other CMI+SMART; 1=DFB Only, DFB+SMART
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would be more likely to participate in at least one session of the BetterChoices, BetterHealth program if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority; p = 0.2211, Regression, Logistic; Odds Ratio (OR) = 0.679, 95% CI 2-sided [0.366 to 1.262] — Modeled probability of attending at least one class. Independent variable coded: 0=Other CMI Only, DFB Only; 1=Other CMI+SMART, DFB+SMART

18. Secondary Outcome: Information Seeking: Use of RA Self-Management Website
Description: The investigators created a website that provided easy access to information about RA, treatment options, and self-management strategies. Participants were emailed a link to this website immediately after completion of 6-week follow-up data collection. The investigators used Google analytics to track whether participants accessed the website.
Time Frame: 6 months
Population: This was an intent to treat analysis. Includes all 265 participants who were given access to the RA Self-Management Website. (Excludes 21 people who withdrew from the study before being given access to this website.)
Measure: Count of Participants; unit: Participants
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 70 | 71 | 63 | 61
Participants
  Visited website at least one time | 13 | 10 | 17 | 10
  Did not visit website | 57 | 61 | 46 | 51
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would be more likely to use the RA Self-Management website if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority; p = 0.5740, Regression, Logistic; Odds Ratio (OR) = 0.804, 95% CI 2-sided [0.38 to 1.72] — Modeled probability of viewing at least one page on website. Independent variable coded: 0=Other CMI Only, Other CMI+SMART, DFB Only; 1=DFB+SMART
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would be more likely to visit the RA Self-Management Website if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority; p = 0.1278, Regression, Logistic; Odds Ratio (OR) = 1.425, 95% CI 2-sided [0.766 to 2.649] — Modeled probability of viewing at least one page on website. Independent variable coded: 0=Other CMI Only, Other CMI+SMART; 1=DFB Only, DFB+SMART
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would be more likely to visit the RA Self-Management Website if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority; p = 0.1278, Regression, Logistic; Odds Ratio (OR) = 0.614, 95% CI 2-sided [0.328 to 1.15] — Modeled probability of viewing at least one page on website. Independent variable coded: 0=Other CMI Only, DFB Only; 1=Other CMI+SMART, DFB+SMART

19. Secondary Outcome: Mean Visual Selective Learning at 6-Month Follow-up Adjusted for Baseline
Description: The Visual Selective Learning (VSL) task will be administered as part of telephone interviews by showing participants 3 lists of 16 words via a PowerPoint presentation embedded in a YouTube video. Each word will appear on a separate screen for 1 second. Half of the words will be in uppercase and half will be in lowercase. In some trials, participants will be instructed that uppercase words are valued at 10 points and lowercase words at 1 point; in other trials, the point value was the opposite. Participants will be told to remember as many words as they could, but that their goal is to earn as many points as possible. Different word lists will be used at each time point and the lists will be balanced across participants over the course of the study using procedures parallel to those for the TOSL. At each time point, scores will be summed across the three lists, yielding a composite score with a possible range from 0 to 264, with higher numbers reflect greater VSL.
Time Frame: Month 6 Follow-up
Population: Includes 224 participants who completed the Visual Selective Learning measure at the 6-month follow-up. (Excludes 62 people who had missing data at the 6-month follow-up.)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 68 | 52 | 60 | 44
score on a scale | 120.1 (6.4) | 109.3 (7.3) | 104.2 (7.6) | 99.2 (8.4)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater increases in visual selective learning between baseline and the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.17, Regression, Linear; Mean Difference (Net) = 11.9, 95% CI 2-sided [-5.2 to 28.9], Standard Error of Mean 8.7 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in visual selective learning between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.02, Regression, Linear; Mean Difference (Net) = 16.0, 95% CI 2-sided [2.5 to 29.5], Standard Error of Mean 6.9 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would experience a greater increase in visual selective learning between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline values of the dependent variable; p = 0.42, Regression, Linear; Mean Difference (Net) = 5.6, 95% CI 2-sided [-8.1 to 19.2], Standard Error of Mean 6.9 — Independent variable coded: 0=Other CMI Only, DFB Only; 1=Other CMI+SMART, DFB+SMART. Difference score calculated as: Comparison Group - Intervention Group. Thus, negative values indicate mean was greater in the intervention group

20. Secondary Outcome: Mean Medication Self-Management Knowledge
Description: Medication Self-Management Knowledge will be assessed using a 45-item medication-specific measure tailored to the medications each participant reports using and developed specifically for this study. The questions will draw on information found in the medication information provided to participants. Correct answers will be summed across the 45 items. Scores transformed to a 100-point scale (ranging from 0-100) with higher values reflecting greater knowledge.
Time Frame: 6 months
Population: Includes 189 participants who had responded to the Medication Self-Management Knowledge items at the 6-month follow-up. (Excludes 97 people who had missing data at the 6-month follow-up.)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 61 | 40 | 51 | 37
score on a scale | 62.4 (1.2) | 64.9 (1.0) | 65.1 (1.1) | 66.1 (1.3)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater medication self-management knowledge at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority; p = 0.15, Regression, Linear; Mean Difference (Net) = -2.2, 95% CI 2-sided [-5.2 to 0.8], Standard Error of Mean 0.15 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit greater medication self-management knowledge at the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority; p = 0.07, Regression, Linear; Mean Difference (Net) = -2.1, 95% CI 2-sided [-4.4 to 0.3], Standard Error of Mean 1.2 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would experience greater medication self-management knowledge at the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority; p = 0.13, Regression, Linear; Mean Difference (Net) = -1.8, 95% CI 2-sided [-4.2 to 0.6], Standard Error of Mean 1.2 — Independent variable coded: 0=Other CMI Only, DFB Only; 1=DFB+SMART, DFB+SMART. Difference score calculated as: Comparison Group - Intervention Group. Thus, negative values indicate mean was greater in the intervention group

21. Secondary Outcome: Mean Verbatim Recall of Information Concerning Medication Benefits and Risks
Description: Verbatim recall of information concerning potential medication benefits and harms will be assessed by medication-specific items developed specifically for this study. For each medication, the investigators will identify one potential benefit and one potential harm listed in the Drug Facts Box. Each question will ask participants about the probability of benefit/harm using a multiple-choice response format. To minimize response burden, participants will be asked these questions in relation to only one of their current RA medications. Correct responses will be summed across the benefit and harm items to yield a score ranging from 0 to 2. Higher numbers reflect greater verbatim recall.
Time Frame: 6 weeks
Population: Includes 190 participants who completed the Verbatim Recall measure at the 6-month follow-up. (Excludes 96 people who had missing data at the 6-month follow-up.)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 62 | 43 | 50 | 35
score on a scale | 0.60 (0.09) | 0.56 (0.10) | 0.44 (0.08) | 0.49 (0.12)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater verbatim recall of information concerning medication benefits and risks at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority; p = 0.68, Regression, Linear; Mean Difference (Net) = 0.05, 95% CI 2-sided [-0.19 to 0.29], Standard Error of Mean 0.12 — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Other CMI Only; The investigators hypothesized that participants would exhibit greater verbatim recall of information concerning medication benefits and risks at the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority; p = 0.20, Regression, Linear; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.06 to 0.31], Standard Error of Mean 0.10 — [estimate comment as in outcome 3, analysis 2]
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would exhibit greater verbatim recall of information concerning medication benefits and risks at the 6-week follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority; p = 0.99, Regression, Linear; Mean Difference (Net) = 0.001, 95% CI 2-sided [-0.19 to 0.19], Standard Error of Mean 0.10 — [estimate comment as in outcome 19, analysis 3]

22. Other Pre Specified Outcome: Patient Interest in Information About Treatment Options: Viewed at Least One Webpage
Description: After participants complete the baseline questionnaire, they were directed to a website that provides written prescription drug information for medications used to treat RA. From baseline to the 6-month follow-up, the investigators electronically tracked the number of webpages viewed and whether participants viewed any of the webpages.
Time Frame: 6 months
Population: This was an intent to treat analysis. Includes all 286 individuals who were given access to the written prescription drug information.
Measure: Count of Participants; unit: Participants
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 78 | 77 | 65 | 66
Participants
  Viewed at least one page | 30 | 18 | 35 | 28
  Did not view any web pages | 48 | 59 | 30 | 38
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would be more likely to view at least one webpage if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority; p = 0.0028, Regression, Logistic; Odds Ratio (OR) = 2.105, 95% CI 2-sided [1.291 to 3.432]; Modeled probability of viewing at least one webpage. Independent variable coded: 0=Other CMI Only, Other CMI+SMART; 1=DFB Only, DFB+SMART

23. Other Pre Specified Outcome: Patient Interest in Information About Treatment Options: Number of Pages Viewed
Description: as for outcome 22
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: pages viewed
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 78 | 77 | 65 | 66
pages viewed | 1.63 (2.8) | 1.39 (4.1) | 2.63 (4.0) | 2.06 (4.0)
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would view more webpages if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority; p = 0.0601, Regression, Linear; Mean Difference (Net) = -0.84, 95% CI 2-sided [-1.71 to 0.04], Standard Error of Mean 0.45 — [estimate comment as in outcome 3, analysis 2]

24. Other Pre Specified Outcome: Percentage of Participants Using a DMARD (Disease-Modifying Antirheumatic Drug) at 6-Month Follow-up
Description: DMARD usage will be assessed via online questionnaires. Participants will be shown a checklist of 19 medications used to treat RA (abatacept, adalimumab, azathioprine, certolizumab pegol, cyclosporine, etanercept, golimumab, gold, hydroxychloroquine, infliximab, leflunomide, methotrexate pill, methotrexate shot, minocycline, rituximab, sulfasalazine, tocilizumab infusion, tocilizumab shot, and tofacitinib) and asked to check all of those that they are currently using. Participants will also be to check an option labeled None of the above. DMARD Usage will be scored as "0" if the participant reports using no DMARDS and "1" if the participant reports using one or more DMARDS.
Time Frame: Month 6 Follow-up
Population: Includes 220 participants who completed the measure assessing medication use at the 6-month follow-up. (Excludes 66 people who had missing data at the 6-month follow-up.)
Measure: Number; unit: percentage of participants
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
Number analyzed (Participants) | 66 | 52 | 59 | 43
percentage of participants
  % Using a DMARD | 93.9 | 86.5 | 93.2 | 93.0
  % Not Using a DMARD | 6.1 | 13.5 | 6.8 | 7.0
Statistical Analysis 1: Comparison: Other CMI Only vs Other CMI & SMART Program vs Drug Facts Boxes Only; The investigators hypothesized that participants would be more likely to be using at least one DMARD (Disease-Modifying Antirheumatic Drug) at the 6-month follow-up if they were assigned to receive medication information via the DrugFactsBox® format combined with gist reasoning training, delivered via the SMART Program, compared to individuals in the other three groups; Test type: Superiority; p = 0.90, Regression, Logistic; Odds Ratio (OR) = 0.91, 95% CI 2-sided [0.22 to 3.81] — Independent variable coded: 0=Other Consumer Medication Information (CMI) Only, Other CMI+SMART, DrugFactsBox® (DFB) Only; 1=DFB+SMART
Statistical Analysis 2: Comparison: Other CMI Only vs Other CMI & SMART Program; The investigators hypothesized that participants would exhibit a greater increase in the percentage of participants using at least one DMARD (Disease-Modifying Antirheumatic Drug) between baseline and the 6-month follow-up if they were assigned to receive written medication information via the DrugFactsBox® format compared to the Other CMI format; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.63, Regression, Logistic; Odds Ratio (OR) = 0.75, 95% CI 2-sided [0.24 to 2.35] — . Independent variable coded: 0=Other Consumer Medication Information (CMI) Only, Other CMI+SMART; 1=DFB Only, DFB+SMART
Statistical Analysis 3: Comparison: Other CMI Only vs Drug Facts Boxes Only; The investigators hypothesized that participants would experience a greater increase in the percentage of participants using at least one DMARD (Disease-Modifying Antirheumatic Drug) between baseline and the 6-month follow-up if they were assigned to receive gist reasoning training, delivered via the SMART Program, compared to those who were not assigned to receive this training; Test type: Superiority — Regression model adjusted for baseline value of the dependent variable; p = 0.81, Regression, Logistic; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.37 to 3.54] — Independent variable coded: 0=Other Consumer Medication Information (CMI) Only, DrugFactsBox® (DFB) Only; 1=Other CMI+SMART, DFB+SMART

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Other CMI Only | Other CMI & SMART Program | Drug Facts Boxes Only | Drug Facts Boxes & SMART Program
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/77 | 0/65 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/77 | 0/65 | 0/66
Other Adverse Events (participants affected / at risk) | 0/78 | 0/77 | 0/65 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT02820038/Prot_SAP_000.pdf